CLINICAL TRIAL: NCT01880476
Title: Feasibility, Acceptability and Effects of an Interprofessional Community-Based Health Promotion Intervention on Self-Management in Older Adults With Type 2 Diabetes and Comorbid Chronic Conditions: A Pilot Study
Brief Title: Interprofessional Community-Based Diabetes Intervention for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Diabetes Care Guelph (Unknown); Guelph Wellington Seniors Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Labarge-13-377
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Comorbidity; Aged; Health Services
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home visits and group program (Experimental)
  Interventions: Other: Home visits and group program

INTERVENTIONS:
Other: Home visits and group program — Participants will receive up to three home visits by a Registered Nurse and two home visits by a Registered Dietitian over the 6-month intervention period. Participants will also be invited to attend a monthly Diabetes Wellness Day group program which will include diabetes education, interaction with peer volunteers, group exercise, and a meal. The Registered Nurse will coordinate care to help participants access necessary community supports and services and lead monthly interprofessional case conferences to develop a client-centred plan of care for each study participant.

SUMMARY:
This study will examine the feasibility and acceptability of a 6-month interprofessional community-based health promotion program, and explore its effects on older adults' self-management of Type 2 Diabetes (T2DM). Recently enrolled clients of Diabetes Care Guelph (DCG), who are age 65+ and have at least two other chronic conditions, will be eligible to participate. Participants must be English speaking, community-dwelling, independent in activities of daily living, and mentally competent to give informed consent. The 6-month intervention will consist of: in-home visits by a Registered Nurse and Registered Dietitian from DCG; participation in a monthly Diabetes Wellness Day group program offered through the Guelph Wellington Seniors Association (GWSA) together with DCG; peer support from trained volunteers at the Diabetes Wellness Day group program; care coordination by the DCG Registered Nurse to help participants access necessary supports and services; and monthly team conferences between care providers at DCG and the GWSA to develop a client-centred plan of care. To evaluate the program, participants will complete interviewer-administered questionnaires before and after the intervention, and care providers and peer volunteers will take part in group interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+
* Referred to Diabetes Care Guelph within the past 12 months
* At least two chronic conditions in addition to Type 2 Diabetes Mellitus
* English speaking
* Community-dwelling, in the city of Guelph
* Independent in activities of daily living
* Mentally competent to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the Summary of Diabetes Self-Care Activities questionnaire | baseline and 6 months
  This questionnaire measures self-care activities including diet, exercise, blood glucose testing, foot care, and smoking.

SECONDARY OUTCOMES:
Changes from baseline in health-related quality of life (SF-12v2 health survey) | Baseline and 6 months
Changes from baseline in depressive symptoms (Centre for Epidemiological Studies Depression Scale) | Baseline and 6 months
Changes from baseline in symptoms of anxiety (Generalized Anxiety Disorder Screener-7 Scale) | Baseline and 6 months
Changes from baseline in costs of use of health services (Health and Social Services Utilization Inventory) | Baseline and 6 months
Changes from baseline in fasting blood glucose (mmol/L) | Baseline and 6 months
Changes from baseline in HbA1C (%) | Baseline and 6 months
Changes from baseline in number of hypoglycemic events per week (blood glucose <4.0 mmol/L) | Baseline and 6 months

OTHER OUTCOMES:
Partnership and collaboration questionnaire | 6 months
  This questionnaire will be completed by care providers who carry out the intervention. It will be used to help evaluate the feasibility and acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, PhD, RN, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Markle-Reid M, Ploeg J, Fisher K, Reimer H, Kaasalainen S, Gafni A, Gruneir A, Kirkconnell R, Marzouk S, Akhtar-Danesh N, Thabane L, Rojas-Fernandez C, Upshur R. The Aging, Community and Health Research Unit-Community Partnership Program for older adults with type 2 diabetes and multiple chronic conditions: a feasibility study. Pilot Feasibility Stud. 2016 May 9;2:24. doi: 10.1186/s40814-016-0063-1. eCollection 2016. PMID 27965843